CLINICAL TRIAL: NCT03279783
Title: LCI (Linked Color Imaging) for Adenoma Detection in the Right Colon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Franco Radaelli, Head of Endoscopy Unit, Valduce Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: 341/2017
Record Dates: First submitted 2017-08-24; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Adenoma Colon Polyp

STUDY DESIGN:
Intervention Model Description: Participants scheduled for colonoscopy for the assessment of symptoms or for colorectal cancer screening/surveillance receive the examination of the right colon twice, in a back-to-back fashion, with standard white light (WL) and with LCI (Linked Color Imaging). Patients are randomly assigned (1:1), via computer-generated randomisation with block size of 20, to which procedure is done first.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WLI (White light Imaging) (No Intervention): Colonoscope withdrawal was performed in the right colon evaluating the mucosa using standard white light.
- LCI (Linked Color Imaging) (Active Comparator): Colonoscope withdrawal was performed in the right colon evaluating the mucosa using LCI (Linked Color Imaging).
  Interventions: Device: LCI (Linked color imaging)

INTERVENTIONS:
Device: LCI (Linked color imaging) — Colonoscope withdrawal was performed in the right colon evaluating the mucosa using LCI (Linked color imaging)
  Arms: LCI (Linked Color Imaging)

SUMMARY:
Although colonoscopy with polypectomy can prevent up to 80% of colorectal cancers, a significant adenoma miss rate still exists, particularly in the right colon. Optimizing the detection of adenomas and sessile serrated lesions in the right colon is crucial to increase the effectiveness of colonoscopy in colorectal cancer prevention.

Last generation Fuji videocolonscopes incorporates the Linked Color Imaging (LCI), a recently developed technology that differentiates the red colour spectrum more effectively than White Light imaging thanks to its optimal pre-process composition of light spectrum and advanced signal processing. The increased colour contrast results in more accurate delineation of abnormal inflammatory or neoplastic findings of colonic mucosa. Preliminary data suggest that LCI may be improve the detection of neoplastic lesion of colon.

The investigators performe a tandem prospective study to compare the right colon adenoma miss rates of LCI colonoscopy with those of conventional white light colonoscopy.

Therefore participants scheduled for colonoscopy for the assessment of symptoms or for colorectal cancer screening/surveillance receive the examination of the right colon twice, in a back to back fashion, with standard white light (WL) and with LCI. Patients are randomly assigned (1:1), via computer-generated randomisation with block size of 20, to which procedure is done first. The endoscopist are masked to group allocation until immediately before the cecum is reached. Examinations are performed with Fuji videocolonscopes series 700 (EC-760R, EC-760ZP).

ELIGIBILITY:
Inclusion Criteria:

* all outpatients referred for colonoscopy

Exclusion Criteria:

* inadequatete bowel preparation (Boston Bowel Preparation Scale (BBPS) < 2 in one colonic segment)
* previous colonic resection
* inflammatory bowel disease
* ereditary polyposic syndromes
* patients on antithrombotics precluding polyp recetion
* absence of informed consent
* inpatients or patients undergoing urgent colonscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Right colon adenoma miss rate | One year
  Number of adenomas identified during the second right coloninspection/ overall number of adenomas identified during the first and the second right colon inspection

SECONDARY OUTCOMES:
Right colon advanced adenomas (size>1 cm and/or high grade displasia and/or villous component) miss rate | One year
  Number of advanced adenomas identified during the second right coloninspection/ overall number of advanced adenomas identified during the first and the second right colon inspection
Right colon sessile serrated lesions miss rate | One year
  Number of sessile serrated lesions identified during the second right coloninspection/ overall number of sessile serrated lesions identified during the first and the second right colon inspection

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Unit, Valduce Hospital, Como, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paggi S, Mogavero G, Amato A, Rondonotti E, Andrealli A, Imperiali G, Lenoci N, Mandelli G, Terreni N, Conforti FS, Conte D, Spinzi G, Radaelli F. Linked color imaging reduces the miss rate of neoplastic lesions in the right colon: a randomized tandem colonoscopy study. Endoscopy. 2018 Apr;50(4):396-402. doi: 10.1055/a-0580-7405. Epub 2018 Mar 14. PMID 29539651